CLINICAL TRIAL: NCT06789367
Title: The Effect of Dexamethasone Administration Route on Pain and Inflammatory Response in PENG Block for Pediatric Hip Surgery
Brief Title: The Effect of Dexamethasone Administration Route in PENG Block for Pediatric Hip Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3/2025
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-01

CONDITIONS: Hip Dysplasia; Hip Disease
Keywords: pericapsular nerve group block; PENG block; dexamethasone; adjuvant
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perinerual dexamethasone (Active Comparator): PENG block + perineural dexamethasone
  Interventions: Drug: perineural Dexamethasone 4mg
- intravenous dexamethasone (Active Comparator): PENG block + intravenous dexamethasone
  Interventions: Drug: intravenous Dexamethsone 4mg

INTERVENTIONS:
Drug: perineural Dexamethasone 4mg — PENG block with 0.5ml/kg 0.2% ropivacaine + 0,1mgkg perineural Dexamethasone
  Arms: perinerual dexamethasone
Drug: intravenous Dexamethsone 4mg — PENG block with 0,5ml/kg 0.2% ropivacaine + 0,1mg/kg intravenous Dexamethasone
  Arms: intravenous dexamethasone

SUMMARY:
This study aims to assess the impact of the administration route of dexamethasone (intravenous vs. perineural) on postoperative pain, inflammatory response, and neuromonitoring parameters in pediatric patients undergoing hip surgery. The primary outcome is postoperative pain intensity measured using an age-appropriate pain scale at multiple time intervals. Secondary outcomes include inflammatory markers such as neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR), opioid consumption, time to first rescue analgesia, and overall patient recovery. This randomized, double-blinded study seeks to improve pain management strategies and optimize anesthesia protocols in pediatric hip surgery.

DETAILED DESCRIPTION:
Pediatric hip surgery is a complex procedure that can result in significant postoperative pain and an inflammatory response. Effective pain management is critical in this population to promote early mobilization, reduce opioid consumption, and minimize adverse outcomes. The pericapsular nerve group (PENG) block is a regional anesthesia technique that offers targeted analgesia for hip procedures while preserving motor function, making it particularly suitable for pediatric patients.

Dexamethasone is commonly used as an adjuvant in regional anesthesia to prolong analgesia and mitigate inflammation. However, the optimal administration route of dexamethasone in the context of PENG block for pediatric hip surgery remains unclear. This study is designed to compare the efficacy of intravenous versus perineural dexamethasone in prolonging postoperative analgesia and reducing inflammatory responses.

This prospective, randomized, double-blinded clinical trial will enroll pediatric patients undergoing elective hip surgery. Participants will be randomized into two groups: one group will receive intravenous dexamethasone, while the other will receive perineural dexamethasone administered as part of the PENG block. All patients will receive standardized general anesthesia and PENG block using a local anesthetic at a fixed concentration.

The primary outcome will be time to first request rescue analgesia. Secondary outcomes include the inflammatory response measured by NLR and PLR, postoperative pain intensity, assessed using an age-appropriate pain scale at predefined time intervals, total opioid consumption, and blood glucose levels. The study will also monitor neuromonitoring parameters during surgery to ensure patient safety and evaluate the influence of dexamethasone on neurological outcomes.

Safety will be closely monitored throughout the study, with particular attention to potential complications such as local anesthetic systemic toxicity (LAST) or dexamethasone-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for hip surgery
* body weight > 5kg

Exclusion Criteria:

* infection at the site of the regional block,
* coagulation disorders,
* immunodeficiency,
* American Society of Anesthesiologists (ASA) physical status of IV or higher,
* history of regular steroid medication.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time to first rescue opioid analgesia

SECONDARY OUTCOMES:
Total opioid consumption | 48 hours after surgery
  Total opioid consumption in milliequivalents of morphine
NRS | 4 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
NRS | 8 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
NRS | 12 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
NRS | 24 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
NRS | 48 hours after surgery
  The numeric rating scale (NRS) with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
Nerve damage | 12 hours after surgery
  Nerve damage assesent will be performed using scale: N0- no nerve damage; N1- minor - sensory paresthesia; N2- majorcomplete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome
Nerve damage | 24 hours after surgery
  Nerve damage assesent will be performed using scale: N0- no nerve damage; N1- minor - sensory paresthesia; N2- majorcomplete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome
Nerve damage | 48 hours after surgery
  Nerve damage assesent will be performed using scale: N0- no nerve damage; N1- minor - sensory paresthesia; N2- majorcomplete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome
NLR | 12 hours after surgery
  Neutrophile-to-lymphocyte ratio
NLR | 24 hours after surgery
  Neutrophile-to-lymphocyte ratio
NLR | 48 hours after surgery
  Neutrophile-to-lymphocyte ratio
PLR | 12 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 24 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymphocyte ratio
glucose | 12 hours after surgery
  blood glucose levels
glucose | 24 hours after surgery
  blood glucose levels
glucose | 48 hours after surgery
  blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, M.D. Ph.D., Study Chair — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes